CLINICAL TRIAL: NCT02735304
Title: Clinical Pilot Study of: Astringent Retraction Paste, Imprint™ 4 VPS, Imprint 4™ Preliminary, Intra-oral Syringes, 3M ESPE New Temporary Restoration (SuPro 100 and Temporary Cement), RelyX™ Unicem™ 2 Automix Cement, Lava™ Plus Zirconia Crowns
Brief Title: Clinical Study 3MESPE Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: 3M ESPE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR15/02 STH 18492
Record Dates: First submitted 2016-03-01; First posted 2016-04-12 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Innovation treatment 3M ESPE materials (Other): The Innovation treatment arm will receive the innovation treatment first and then crossover to receive the standard clinical practice treatment during the Impression intervention.
  Materials to be used all 3M ESPE - Astringent Retraction Paste, Imprint™ 4 Preliminary, Imprint™4 VPS, Imprint™ 4 Bite, Intra-oral syringes, Impression Tray,
  Interventions: Other: Impression intervention
- standard clinical practice treatment (Other): The standard clinical practice treatment will receive the standard clinical practice treatment first and then crossover to receive the innovation treatment during the Impression intervention
  Materials as per the operating dentist's choice to be recorded on CRF
  Interventions: Other: Impression intervention

INTERVENTIONS:
Other: Impression intervention — The 1st intervention will compare two clinical impression techniques The Innovation treatment arm will receive the innovation treatment first and then crossover to receive the standard clinical practice treatment. The standard clinical practice treatment will receive the standard clinical practice treatment first and then crossover to receive the innovation treatment.

SUMMARY:
This clinical study seeks to address four independent questions that are all part of the delivery of care associated with the provision of a single item of treatment; an indirect restoration (known as a 'crown') to restore and cover a damaged tooth. The provision of a crown requires a series of sequential clinical and laboratory stages stages:

1. Stage 1 - Preliminary impression. Taking a pre-operative impression of the tooth to be crowned. This will be used to enable the fabrication of the temporary crown after the tooth has been prepared. This is standard care and follows established clinical protocols.
2. Stage 2 - Preparation of the tooth. This involves cutting the tooth back to make space for the crown that will be fabricated to replace the missing structure.
3. Stage 3 - Taking an impression of the prepared tooth. From this a duplicate model will be made to fabricate the crown. To take the impression, the dentist will need to gently push the gums away from the tooth by fractions of a millimeter so that the margins of the preparation are clearly discernible.
4. Stage 4 - Provision of a temporary restoration that will provide satisfactory function for a limited period of time, until the definitive crown can be fitted. This temporary crown is designed to have a finite short-term durability and have an ease of manufacture and subsequent removal; hence the use of a specific cement that will enable this.
5. Stage 5 - Fitting of the definitive restoration. This is designed to be a durable restoration, with a mean life expectancy measured in years, but which is ultimately determined by a number of clinical, biological and patient specific parameters. Definitive restorations are fitted with cement designed to retain the crown in permanent manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of at least one full-coverage posterior restoration (crown) in a permanent premolar or molar.
* If two teeth in opposing arches are in need of a full-coverage posterior restoration (crown) only the tooth or teeth in one arch will be included in the study.

Exclusion Criteria:

* Patients who are unable to give informed consent or vulnerable population as defined in ISO 14155 will not be enrolled.
* Patients with contraindications as described in the 'Instructions for Use' of the study materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the predictability | 48 months
  Assessment of the predictability of results as a function of accuracy of the resulting model, the dentist's judgment on the quality of impression and the accuracy of fit of the definitive restoration (Lava™ Plus Zirconia crown). Predictability is defined as the frequency in which an adequate result is obtained in a consistent manner

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martin, Professor, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Sheffield NHS Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plans to share data